CLINICAL TRIAL: NCT01483391
Title: Early Intervention for Youth at Risk for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Stanford University (Other); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH093676 (NIH)
Record Dates: First submitted 2011-11-26; First posted 2011-12-01 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
Keywords: Bipolar disorder; Major depressive disorder; Mania; Depression; Cyclothymic Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Mania; Depression; Cyclothymic Disorder | interventions — Case Management; Family Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Care (Active Comparator): Three sessions of family education and three sessions of individual support over 4 months.
  Interventions: Behavioral: Enhanced Care
- Family-Focused Treatment (Experimental): 12 therapy sessions involving the at-risk child or adolescent, parents, and available siblings. Therapy will include psychoeducation about mood disorders, communication enhancement training, and problem-solving skills training.
  Interventions: Behavioral: Family-Focused Treatment

INTERVENTIONS:
Behavioral: Enhanced Care — The 3 family sessions involve the youth and all family members. These sessions will help the child and family members with mood charting and developing a mood management plan. Families will rehearse mood regulation strategies for current family, social or academic problems. Clinicians then meet with the child individually every month for the next 3 mos. to provide support, assist with problem-solving, and troubleshoot use of the mood management plan.
  Other Names: Psychoeducation; Case Management
  Arms: Enhanced Care
Behavioral: Family-Focused Treatment — 12 therapy sessions involving the at-risk child or adolescent, parents, and available siblings. Therapy will include psychoeducation about mood disorders, communication enhancement training, and problem-solving skills training. The goal of this intervention is to improve the child's ability to regulate moods and to reduce tension and conflict in the family.
  Other Names: Family Therapy; Family Psychoeducation; FFT; Family Intervention; Psychoeducation; Family Treatment
  Arms: Family-Focused Treatment

SUMMARY:
Children or teens with mood swings or depression who have a parent with bipolar disorder are at high risk for developing bipolar disorder themselves. This study will test a family-based therapy aimed at preventing or reducing the early symptoms of bipolar disorder in high-risk children (ages 9-17). In a randomized trial, the investigators will compare two kinds of family-based treatment (one more and one less intensive) on the course of early mood symptoms and social functioning among high-risk children followed for up to 4 years. The investigators will examine the effects of family treatment on measures of neural activation using functional magnetic resonance imaging.

DETAILED DESCRIPTION:
Children who are at high risk for developing bipolar disorder (BD) often are showing significant mood swings or depression well before they develop the full disorder. Often, these children have one or more parents who have bipolar disorder. In addition to brief episodes of lethargic depression and mania or hypomania (periods of excessive activity), children and adolescents at risk for BD often have co-occurring disorders, such as attention deficit hyperactivity disorder, conduct disorder, substance abuse disorders, and anxiety disorders.

Early interventions may lead to better mental health by preventing BD from ever fully expressing itself. This study will test an early intervention for BD called family-focused treatment (FFT), which has been designed to help children and adolescents who are at risk for developing BD. FFT will combine education about BD with training in communication strategies and problem-solving skills. It will focus on the family, because family environmental factors are related to the course and recurrence of BD. By reducing risk factors and teaching coping skills, FFT aims to reduce the early symptoms of BD, improve functioning, and delay the onset or reduce the severity of manic episodes.

Participation in this study will last up to 4 years, although the majority of the study will occur in the first year. There are three parts. In the first part, participating children and their families will complete research interviews and questionnaires about the child's mood, behavior, beliefs, and problems. Parent participants will provide information on the family background of mood or anxiety problems. All participants will receive a thorough medical-psychiatric evaluation and be provided with pharmacotherapy (as needed) from a study psychiatrist for the first year of the study.

In the second part, participants will be randomly assigned to receive one of two treatments: FFT or enhanced care. Participants receiving FFT will complete 12 therapy sessions in which parents, children, and siblings learn how to cope with mood disorders, new ways to talk to each other, and strategies for solving family problems. FFT sessions will occur weekly for the first 8 weeks and then every other week for the next 8 weeks. Participants receiving enhanced care will have 3 weekly sessions which will involve the youth and all family members. In session 1, clinicians summarize the diagnostic assessment, introduce mood charting, and offer instructional handouts on managing mood swings. In session 2, clinicians revisit mood charting, discuss medications (if relevant), and help the child and family develop a mood management plan. In session 3, families rehearse mood regulation strategies for current family, social or academic problems. Clinicians then meet with the child individually every month for the next 3 mos. to provide support, assist with problem-solving, and troubleshoot use of the mood management plan. So, both treatments last 4 months.

In the third part of the study, participants will complete follow-up assessments every 4 months for 1 year. Assessments will include interviews and questionnaires similar to those completed in the first part of the study.

The statistical analyses for this study will examine changes in symptoms and functioning from the baseline assessment through the 4 month follow-ups in year 1 and the 6 month follow-ups in years 2-4.

ELIGIBILITY:
Inclusion Criteria:

* For a child to be eligible:

  * At least one biological parent or stepparent with whom the child or adolescent lives must be willing to participate in family treatment
  * At least one biological parent has a verifiable diagnosis of bipolar disorder I or II
  * The child must have a DSM-IV diagnosis of bipolar disorder not otherwise specified or major depressive disorder (MDD)
  * If the main diagnosis is MDD, the depressive episode must have occurred within the past 2 years
  * The child must have evidence of current significant affective symptoms, as determined by a score greater than 11 on the Young Mania Rating Scale within the last week or a score greater than 29 on the Child Depression Rating Scale-Revised within the last 2 weeks
  * The family must speak English, although English need not be their first language

Exclusion Criteria:

* Fully diagnosable bipolar disorder I or II
* Diagnosis of autism or pervasive developmental disorder
* Evidence of mental retardation, as defined by an intelligence quotient (IQ) less than 70
* Presence of comorbid neurologic diseases such as seizure disorder
* Substance or alcohol abuse or dependence disorders in the 4 months prior to study recruitment
* Evidence of a life-threatening eating disorder or other medical disorder that requires emergency medical treatment
* Currently enrolled in regular family therapy
* Evidence of current sexual or physical abuse or domestic abuse between the adult partners

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2011-10-06 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in symptom severity | Measured at baseline, every 4 months in year 1, and every 6 months in years 2-4
  Changes in symptoms of at-risk children, as defined by depression and (hypo)mania scores and psychiatric status on the Adolescent Longitudinal Interval Follow-up Evaluation (A-LIFE, the Child Depression Rating Scale, and the Young Mania Rating Scale

SECONDARY OUTCOMES:
Delaying onset of a first (hypo)manic or mixed episode | 2-4 years
  We will evaluate through survival analyses whether family-focused treatment, due to its ameliorative effects on acute symptoms, is superior to enhanced care in delaying onset of a first (hypo)manic or mixed episode during the 2-4 year follow-up.
Psychosocial functioning | Measured at baseline, every 4 months in year 1 and every 6 months in years 2-4
  Youths in family-focused treatment will show greater improvement from pretreatment to end of a 2-4 year follow-up in psychosocial functioning compared to youth in Enhanced Care.
Mental health service use | Measured at baseline, every 4 months in year 1 and every 6 months in years 2-4
  Youth in family-focused treatment will require fewer mental health services from pretreatment to end of a 2-4 year follow-up than youth in enhanced care

CONTACTS AND LOCATIONS:
Overall Officials: David J Miklowitz, PhD, Principal Investigator — UCLA Department of Psychiatry; Kiki D Chang, MD, Principal Investigator — Stanford University; Christopher D Schneck, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - UCLA Child and Adolescent Mood Disorders Program, UCLA School of Medicine, Los Angeles, California
  - Stanford University School of Medicine, Lucile Packard Children's Hospital, Stanford, California
  - University of Colorado, Boulder, Boulder, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Upon completing the study we will submit a CD-ROM to the NIH Freedom of Information Act Coordinator containing all raw data, variable coding information, and copies of measures. Prior to archiving the data, we will remove all personal identifiers and other protected information. The youth's and parents' consent forms will make clear that the data, minus any identifying information, will be made available to other researchers at the end of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 1/01/21-1/01/23

REFERENCES:
- [Background] Miklowitz DJ, Chang KD. Prevention of bipolar disorder in at-risk children: theoretical assumptions and empirical foundations. Dev Psychopathol. 2008 Summer;20(3):881-97. doi: 10.1017/S0954579408000424. PMID 18606036
- [Background] Miklowitz DJ, Chang KD, Taylor DO, George EL, Singh MK, Schneck CD, Dickinson LM, Howe ME, Garber J. Early psychosocial intervention for youth at risk for bipolar I or II disorder: a one-year treatment development trial. Bipolar Disord. 2011 Feb;13(1):67-75. doi: 10.1111/j.1399-5618.2011.00890.x. PMID 21320254
- [Derived] Miklowitz DJ, Weintraub MJ, Singh MK, Walshaw PD, Merranko JA, Birmaher B, Chang KD, Schneck CD. Mood Instability in Youth at High Risk for Bipolar Disorder. J Am Acad Child Adolesc Psychiatry. 2022 Oct;61(10):1285-1295. doi: 10.1016/j.jaac.2022.03.009. Epub 2022 Mar 17. PMID 35307538
- [Derived] Singh MK, Nimarko AF, Garrett AS, Gorelik AJ, Roybal DJ, Walshaw PD, Chang KD, Miklowitz DJ. Changes in Intrinsic Brain Connectivity in Family-Focused Therapy Versus Standard Psychoeducation Among Youths at High Risk for Bipolar Disorder. J Am Acad Child Adolesc Psychiatry. 2021 Apr;60(4):458-469. doi: 10.1016/j.jaac.2020.07.892. Epub 2020 Aug 1. PMID 32745598
- [Derived] Miklowitz DJ, Schneck CD, Walshaw PD, Singh MK, Sullivan AE, Suddath RL, Forgey Borlik M, Sugar CA, Chang KD. Effects of Family-Focused Therapy vs Enhanced Usual Care for Symptomatic Youths at High Risk for Bipolar Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):455-463. doi: 10.1001/jamapsychiatry.2019.4520. PMID 31940011
- [Derived] Miklowitz DJ, Portnoff LC, Armstrong CC, Keenan-Miller D, Breen EC, Muscatell KA, Eisenberger NI, Irwin MR. Inflammatory cytokines and nuclear factor-kappa B activation in adolescents with bipolar and major depressive disorders. Psychiatry Res. 2016 Jul 30;241:315-22. doi: 10.1016/j.psychres.2016.04.120. Epub 2016 May 7. PMID 27227701
- See also: UCLA Child and Adolescent Mood Disorders Program — http://www.semel.ucla.edu/champ
- See also: Stanford University Pediatric Bipolar Disorders Program — https://med.stanford.edu/childpsychiatry/clinical/bipolar.html
- See also: University of Colorado Depression Center — http://www.coloradodepressioncenter.org